CLINICAL TRIAL: NCT04453189
Title: A Phase 1, Open-label, Randomized, 2-Way Crossover Study to Assess the Effects of Acid-Reducing Agent(s) on the Pharmacokinetics of a Single Oral Dose of JNJ-64417184 in Healthy Adult Participants
Brief Title: A Study to Assess the Effects of Acid-Reducing Agent(s) on JNJ-64417184 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108812; 2020-000380-23 (EudraCT Number); 64417184RSV1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Lansoprazole; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Sequence: AB(Part 1) followed by C(Part 2-Optional) (Experimental): Participants will received Treatment A (single dose of JNJ-64417184 in fed condition on Day 1) in period 1 followed by Treatment B (lansoprazole on Day 1 to 4 under fasted condition and 2 hours before single dose of JNJ-64417184 in fed condition on Day 5) in period 2 of part 1. There will be a washout period of 7 days between each treatment. Participants will receive Treatment C: optional (famotidine under fasted conditions administered 12 hours before and 12 hours after a single dose of JNJ-64417184 under fed conditions on Day 1) in Part 2, Period 3.
  Interventions: Drug: JNJ-64417184; Drug: Lansoprazole; Drug: Famotidine
- Treatment Sequence: BA(Part 1) followed by C(Part 2-Optional) (Experimental): Participants will receive Treatment B in period 1 followed by Treatment A in period 2, Part 1. There will be a washout period of 7 days between each treatment. Participants will receive Treatment C: optional (famotidine under fasted conditions administered 12 hours before and 12 hours after a single dose of JNJ-64417184 under fed conditions on Day 1) in Part 2, Period 3.
  Interventions: Drug: JNJ-64417184; Drug: Lansoprazole; Drug: Famotidine

INTERVENTIONS:
Drug: JNJ-64417184 — Participants will receive single dose of JNJ-64417184 in fed condition on Day 1 in assigned treatment sequence.
Drug: Lansoprazole — Participants will receive lansoprazole once daily in fasted condition on Day 1 to 4 under fasted condition and 2 hours before single dose of JNJ-64417184 in fed condition on Day 5 in assigned treatment sequence.
Drug: Famotidine — Participant will receive famotidine in fasted condition on Day 1 in assigned treatment sequence.

SUMMARY:
The primary purpose of this study is to evaluate the effect of multiple-dose administration of lansoprazole on the single-dose pharmacokinetics (PK) of JNJ-64417184 in healthy adult participants; and to evaluate the effect of time-separated, multiple-dose administration of famotidine on the single-dose PK of JNJ-64417184 in healthy adult participants (optional).

ELIGIBILITY:
Inclusion Criteria:

* Must have a body mass index (BMI) between 18.0 and 30.0 kilograms per square meters [kg/m^2]), extremes included, and body weight not less than 50.0 kilograms (kg) at screening
* Healthy on the basis of physical examination, medical and surgical history, and vital signs performed at screening
* Healthy on the basis of clinical laboratory tests performed at screening
* Must have a normal 12-lead Electrocardiogram (ECG) (triplicate) at screening, including: normal sinus rhythm (heart rate between 45 and 100 beats per minute [bpm], extremes included); QT interval corrected for heart rate (QTc) according to Fridericia (QTcF) less than or equal to (<=) 450 milliseconds (ms) for male participants and <= 470 ms for female participants; QRS interval less than (<) 120 ms; PR interval <= 200 ms. If the results of the ECG are outside the normal ranges, the participant may be included only if the investigator judges the deviations from normal ECG to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Must sign an informed consent form (ICF) indicating he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study, before starting any screening activities

Exclusion Criteria:

* History of liver or renal dysfunction (calculated creatinine clearance/estimated glomerular filtration rate (eGFR) <60 milliliter per minute (mL/min) at screening, calculated by the Modification of Diet in Renal Disease [MDRD] formula), significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* Past history of clinically significant cardiac arrhythmias (for example, extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (for example, hypokalemia, family history of long QT Syndrome)
* Any evidence of clinically significant heart block or bundle branch block at screening
* Current human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at screening
* History of hepatitis A, B, or C infection, or current hepatitis A infection (confirmed by hepatitis A antibody immunoglobulin M [IgM]), or hepatitis B virus (HBV) infection (confirmed by hepatitis B surface antigen), or HCV infection (confirmed by hepatitis C virus [HCV] antibody) at screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Analyte Concentration (Cmax) of JNJ-64417184 | Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 36, 48, 72, 96, 120 hours and up to follow-up 1 (up to 120 hours in case of dropout; at the time of dropout or the following morning)
  Cmax is defined as the maximum observed plasma analyte concentration.
Area Under the Plasma Analyte Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration (AUC[0-last]) of JNJ-64417184 | Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 36, 48, 72, 96, 120 hours and up to follow-up 1 (up to 120 hours in case of dropout; at the time of dropout or the following morning)
  AUC(0-last) is defined as the area under the plasma analyte concentration-time curve from time 0 to time of the last quantifiable (non-below quantification limit [non-BQL]) concentration calculated by linear-linear trapezoidal summation.
Area Under the Plasma Analyte Concentration-time Curve From Time 0 to Infinite Time (AUC[0-infinity]) of JNJ-64417184 | Predose, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 36, 48, 72, 96, 120 hours and up to follow-up 1 (up to 120 hours in case of dropout; at the time of dropout or the following morning)
  Area under the plasma analyte concentration-time curve from time 0 to infinite time, calculated as AUC (0-last) + C (0-last)/lambda(z), where C (0-last) is the last observed measurable (non BQL) plasma analyte concentration; AUC (0-last) is the area under the plasma analyte concentration-time curve from time 0 to time of the last quantifiable (non-below quantification limit [non-BQL]) concentration and lambda(z) is the terminal phase rate constant. Extrapolations of more than 20.00 percent (%) of the total AUC are reported as approximations.

SECONDARY OUTCOMES:
Number of Participants with Adverse Event as a Measure of Safety and Tolerability | Up to 2.5 months
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.
Number of Participants with Clinically Significant Changes in Vital Signs | Up to 2.5 years
  Number of participants with clinically significant abnormalities in vital signs (Systolic and diastolic blood pressure and pulse rate) will be assessed.
Number of Participants with Clinically Significant Abnormalities in Laboratory Parameters | Up to 2.5 years
  Number of participants with clinically significant abnormalities in laboratory parameters (Hematology Panel, biochemistry panel, coagulation and urinalysis) will be assessed.
Number of Participants with Clinically Significant Abnormalities in Electrocardiogram | Up to 2.5 years
  Number of participants with clinically significant abnormalities in electrocardiogram will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency